CLINICAL TRIAL: NCT05554666
Title: A Phase 1 Dose Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ASKG315 as a Single Agent in Patients With Locally Advanced or Metastatic Malignant Solid Tumors.
Brief Title: A Study of ASKG315 in Patients With Advanced Solid Tumors.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AskGene Pharma, Inc. (Industry)
Collaborators: Jiangsu Aosaikang Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASKG315-001
Record Dates: First submitted 2022-09-19; First posted 2022-09-26 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2022-09

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASKG315 (Experimental): Single or multiple ascending dose of ASKG315
  Interventions: Biological: ASKG315

INTERVENTIONS:
Biological: ASKG315 — Injection with dose escalation stage of 3mg up to 45mg as well as dose expansion stage with recommended dose level from dose escalation stage.

SUMMARY:
The study is a Phase 1, open-label, multicenter, dose escalation study to evaluate the safety, tolerability, PK and PD of ASKG315 as a single agent in patients with advanced solid tumors.

DETAILED DESCRIPTION:
Each part of the study consists of 3 periods: screening (up to 28 days), treatment and follow-up. After an initial screening period, ASKG315 will be administered once every 3 weeks by intravenous (IV) infusion. The Part 1 dose escalation consists of 6 planned escalation cohorts, with a starting dose of 3 mg.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age.
2. Histologically or cytologically confirmed advanced malignant solid tumor that is refractory to or intolerant of all standard therapy or for which no standard therapy is available.
3. Measurable disease, per RECIST v1.1.
4. ECOG Performance Status of ≤ 2.
5. Life expectancy of ≥3 months, in the opinion of the Investigator.
6. Adequate organ function defined.
7. Fertile patients must be willing to use effective contraceptive measures (hormonal or barrier methods or abstinence, etc.) during the trial and at least 90 days after the last dose;negative serum pregnancy test for female patients within 7 days prior to the first dose of the study drug or documentation of lack of childbearing potential.
8. Voluntarily enrolled and signed the informed consent form, followed the experimental treatment plan and visit arrangement.

Exclusion Criteria:

1. Received chemotherapy within 3 weeks prior to Cycle 1 Day 1; received radiotherapy, biotherapy, endocrine therapy, targeted therapy, immunotherapy, or any other anti-tumor treatments within 4 weeks prior to Cycle 1 Day 1.
2. Received any other investigational drug for treatment that is not commercially available within 4 weeks prior to Cycle 1 Day 1.
3. Had major organ surgery or significant trauma within 4 weeks prior to C1D1 or planning elective surgery during the study period.
4. Received systemic glucocorticoid or other immunosuppressant treatment within 2 weeks prior to C1D1.
5. Received immunomodulatory drugs, including but not limited to thymosin and interferon, within 2 weeks prior to C1D1.
6. Received a live attenuated vaccine within 4 weeks prior to C1D1.
7. Received IL-2 or IL-15 therapy within 4 weeks prior to C1D1.
8. History of hematologic stem cell transplant or solid organ transplant.
9. Adverse reactions to previous antitumor therapy have not recovered to CTCAE 5.0 grade ≤ 1.
10. Cerebral parenchymal metastasis or meningeal metastasis with clinical symptoms.
11. Serious infection requiring intravenous infusion or hospitalization, or active viral infection.
12. Current clinically significant interstitial lung disease.
13. History of serious cardiovascular or cerebrovascular diseases.
14. Active or recurrent autoimmune diseases.
15. History of Grade ≥ 3 Immune-Related Adverse Events (irAE) or Grade ≥ 2 immunotherapy-associated myocarditis associated.
16. Other malignancies within 5 years.
17. Bleeding symptoms of CTCAE 5.0 grade ≥3 within 4 weeks prior to C1D1.
18. Symptomatic with uncontrolled ascites or pleural effusion.
19. Hyperglycemia that cannot be stably controlled.
20. History of a grade ≥ 3 allergic reaction to protein drugs.
21. Known to have alcohol or drug dependence.
22. Severe mental disorder or poor compliance.
23. Pregnant or nursing women
24. Subjects should be excluded in the opinion of investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLTs) | 21days
  To evaluate the safery of ASKG315 in subjects.
Adverse events(AEs) | 21days
  To evaluate the safery of ASKG315 in subjects.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | 21days
  To evaluate the systemic pharmacokinetics of ASKG315 in subjects.
Area under the concentration time curve (AUC) | 21days
  To evaluate the systemic pharmacokinetics of ASKG315 in subjects.
Cytokine | 21days
  Increase in circulating cytokine levels.
Immunocyte | 21days
  Changes in immunocyte levels by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, MD, Principal Investigator — Shanghai East Hospital
Locations (4):
- China (4):
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - the First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shandong cancer hospital, Jinan, Shandong
  - Shanghai East Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD or supporting information available.